CLINICAL TRIAL: NCT02766088
Title: A Cohort Study to Assess the Burden of Dengue Illness in Household Members From Selected Communities in Southeast Asia and Latin America
Brief Title: This Study Will Describe the Burden of DENgue Fever Virus (DENV) Illness Among Household Members Aged 6 Months to 50 Years of Selected Communities in Latin America and Southeast Asia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200318
Record Dates: First submitted 2016-04-14; First posted 2016-05-09 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Dengue; Dengue Vaccines
Keywords: Dengue; Household; Southeast Asia; Latin America; Surveillance
MeSH Terms: conditions — Dengue

ARMS (1):
- Total Group (Experimental): Subjects aged between 6 months and 50 years at the time of enrolment living in geographically-defined communities in Latin America and Southeast Asia. The study population comprised household members and should include between 30% and 50% of adults (aged 18 years or above) per site.The appropriate recruitment strategy was selected by each participating site. Two approaches might be considered: a school-based approach and a community-based approach without school involvement The expected period for recruiting the target sample size was approximately three months.
  Interventions: Procedure: Blood sample collection

INTERVENTIONS:
Procedure: Blood sample collection — All participants will have an enrolment visit with collection of a blood sample and a termination contact/visit. Participants or their parents/guardians will be contacted weekly or every two weeks to monitor the occurrence of febrile episodes. Additional visits will be made if febrile episodes occur. In case of dengue suspicion, a blood sample will be collected.

SUMMARY:
The purpose of this study is to describe the burden of DENV illness among household members aged 6 months to 50 years of selected communities in Latin America and Southeast Asia.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent (and assent if the subject is below the legal age of consent) obtained from the subject/from subject's parent(s)/LAR(s). For a subject below the legal age of consent is, his/her signature will be obtained on the informed assent form, if applicable.
* A male or female between, and including 6 months and 50 years of age at the time of enrolment (Subjects become ineligible on their 51st birthday).
* Subject and/or the subject's parent(s)/LAR(s) who the investigator believes can comply with the requirements of the protocol (e.g., willingness to go to the hospital/healthcare centre for visit(s) in case of acute febrile illness, able to observe the signs of dengue and to understand how to take and report body temperature, etc).
* Subject who plans, at the time of enrolment, to remain at same residence/study area during the one or two year study period (as applicable).
* Household should be reachable by phone (residence phone or mobile phone). Note: Pregnant or lactating female or female planning to become pregnant can be recruited into the study.

Exclusion Criteria:

* Child in care.
* Participation (current or planned) in another epidemiological study or in a clinical trial that would conflict with the current study, based on investigator's judgement.
* Terminal illness or severe mental incapacity.

Ages: 6 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1750 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (2):
- GSK Investigational Site, Zapopan, Jalisco, Mexico
- GSK Investigational Site, City of Muntinlupa, Philippines

REFERENCES:
- [Background] DeAntonio R, Amaya-Tapia G, Ibarra-Nieto G, Huerta G, Damaso S, Guignard A, de Boer M. Incidence of dengue illness in Mexican people aged 6 months to 50 years old: A prospective cohort study conducted in Jalisco. PLoS One. 2021 May 5;16(5):e0250253. doi: 10.1371/journal.pone.0250253. eCollection 2021. PMID 33951076
- [Background] Capeding MR, de Boer M, Damaso S, Guignard A. Assessing the burden of dengue among household members in Alaminos, Laguna, the Philippines: a prospective cohort study. Asian Biomed (Res Rev News). 2021 Oct 29;15(5):213-222. doi: 10.2478/abm-2021-0027. eCollection 2021 Oct. PMID 37551324

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In December 2017, GSK decided to deprioritize the development of the dengue purified inactivated vaccine (DPIV) candidate. This decision was made due to the significant scientific challenges of dengue vaccine development. Hence, only 2 sites participated to the study, 1 in Mexico and 1 in Philippines.
Groups:
- Total Group: Subjects aged between 6 months and 50 years at the time of enrolment living in geographically-defined communities in Latin America and Southeast Asia. The study population comprised household members and should include between 30% and 50% of adults (aged 18 years or above) per site.The appropriate recruitment strategy was selected by each participating site. Two approaches were considered: a school-based approach and a community-based approach without school involvement The expected period for recruiting the target sample size was approximately three months.
Period: Overall Study
Arm/Group | Total Group
Started | 850
Completed | 344
Not Completed | 506
Not completed — Sponsor study termination | 498
Not completed — Migrated/moved from the study area | 1
Not completed — Lost to Follow-up | 5
Not completed — Other | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Total Group
Number analyzed (Participants) | 850
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.4 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 456
  Male | 394
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Percentage of Reverse Transcriptase Quantitative Polymerase Chain Reaction (RT-qPCR) Confirmed Symptomatic Dengue Infection During the Study Period by Study Site
Description: Incidence percentage of RT-qPCR confirmed symptomatic dengue infection was expressed as percentage of subjects = (n [number of subjects with at least one event reported during the study period ]/N [number of subjects in the population]) X 100. The 95% Wald CI was calculated. Clustering effect was not retained because equal or less than 1. RT-qPCR confirmed symptomatic case = suspected dengue case (SDC) confirmed by RT-qPCR. See SDC definition in outcome 5.
Time Frame: From Day 0 to Month 24 (study end)
Population: Analysis was performed on the According-to-Protocol cohort that included all evaluable subjects, i.e. subjects who met all eligibility criteria, complying with the procedures defined in the protocol and for whom data of at least one follow-up contact were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 850
Percentage of subjects
  Mexico: number analyzed (Participants) | 350
  Mexico | 1.1 [0.4 to 3.0]
  Philippines: number analyzed (Participants) | 500
  Philippines | 0.8 [0.3 to 2.1]

2. Secondary Outcome: Number of Subjects With DENV-type Specific Confirmed Symptomatic DENV Infection
Description: Dengue Virus (DENV)-Type 1, 2 3 or 4 Ribonucleid acid would have been considered for this analysis but it was not performed due to the low number of cases reported.
Time Frame: From Day 0 to Month 24 (study end)
Population: No data was collected by DENV-type due to the low number of cases reported, therefore no analysis could be performed.
Arm/Group | Total Group
Number analyzed (Participants) | 0

3. Secondary Outcome: Incidence Proportion of Virologically Confirmed Symptomatic Dengue Infection During the Study Period in Mexico
Description: Incidence proportion of virologically confirmed symptomatic dengue infection was estimated from GEE logistic regression model taking the clustering effect into account. The 95% confidence interval was based on the robust variance estimate from the GEE model. Clusters were households for analysis by study site. Virologically confirmed symptomatic case = suspected dengue case (SDC) confirmed by RT-qPCR or non-structural protein 1 (NS1). See SDC definition in outcome 5.
Time Frame: From Day 0 to Month 24 (study end)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 350
Proportion of subjects | 1.4 [0.5 to 3.8]

4. Secondary Outcome: Incidence Percentage of Virologically Confirmed Symptomatic Dengue Infection During the Study Period in the Philippines.
Description: Incidence percentage of virologically confirmed symptomatic dengue infection was expressed as percentage of subjects = (n [number of subjects with at least one event reported during the study period]/N [number of subjects in the population]) X 100. The 95% Wald CI was calculated. Clustering effect was not retained because equal or less than 1. RT-qPCR confirmed symptomatic case = suspected dengue case (SDC) confirmed by RT-qPCR. See SDC definition in outcome 5.
Time Frame: From Day 0 to Month 24 (study end)
Population: Analysis was performed on the According-to-Protocol cohort that included all evaluable subjects from the Philippines, i.e. subjects who met all eligibility criteria, complying with the procedures defined in the protocol and for whom data of at least one follow-up contact were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 500
Percentage of subjects | 0.8 [0.3 to 2.1]

5. Secondary Outcome: Incidence Proportion of Probable Symptomatic Dengue Infection During the Study Period.
Description: Incidence proportion of probable confirmed symptomatic dengue infection was estimated from GEE model with clustering effect. Clusters were households for analysis by study site and study sites for analysis on overall study sites. A probable confirmed dengue infection is an SDC with DENV RT-qPCR negative or not performed (late presenter), and DENV NS1 negative or undetermined (early or late presenter), and Anti-DENV Immunoglobulin type M (IgM) positive with a rapid immunochromatographic (ICT) assay or an Enzyme-linked Immunosorbent Assay (ELISA) assay, or Anti-DENV IgG positive (rapid ICT assay or 'capture ELISA' assay). SDC defined as acute febrile illness measured as greater or equal to 38.0°C or recent history of febrile illness (onset in the past 8 days) reported for at least 2 consecutive days (duration of approximately 36-48 hours) and < 7 days duration, which might be accompanied by other dengue symptoms or signs with no defined focus or obvious reason unrelated to dengue.
Time Frame: From Day 0 to Month 24 (study end)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 850
Proportion of subjects | 0 [NA to NA] — The 95% CI was not calculated as no cases reported.

6. Secondary Outcome: Proportion of Subjects With Dengue Virus Antibody IgG Positive Result (ELISA) at First Visit (Indicative of Past DENV Infection), by Study Site and Age Category.
Description: The proportion of subjects with Dengue Virus antibody IgG positive result (ELISA) was estimated from GEE model with clustering effect. The 95% CI was based on the robust variance estimate from the GEE model. Clusters were households for analysis by study site. Ages categories were defined as follows: "6 months -<12 Months" = from the 6 Months birthday up to and including the day before the 1st year birthday, and the next "n-p Years" categories = from the nth Year birthday up to and including the day before the (p+1)th Year birthday. Analysis was not summarized for confirmed and probable dengue cases, separately, as there were no probable cases reported in the study.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 782
Proportion of subjects
  Mexico- 6 months -12 months: number analyzed (Participants) | 2
  Mexico- 6 months -12 months | 0 [NA to NA] — The 95% CI was not calculated as no cases reported.
  Mexico- 5-8 years: number analyzed (Participants) | 43
  Mexico- 5-8 years | 11.8 [4.5 to 27.5]
  Mexico- 9-17 years: number analyzed (Participants) | 95
  Mexico- 9-17 years | 16.6 [9.8 to 26.6]
  Mexico- 18-50 years: number analyzed (Participants) | 160
  Mexico- 18-50 years | 27.2 [19.8 to 36.2]
  Philippines- 1-4 years: number analyzed (Participants) | 74
  Philippines- 1-4 years | 31.2 [21.7 to 42.7]
  Philippines- 5-8 years: number analyzed (Participants) | 85
  Philippines- 5-8 years | 51.5 [40.8 to 62.0]
  Philippines- 9-17 years: number analyzed (Participants) | 173
  Philippines- 9-17 years | 92.0 [86.4 to 95.4]
  Philippines- 18-50 years: number analyzed (Participants) | 150
  Philippines- 18-50 years | 99.3 [95.4 to 99.9]

7. Secondary Outcome: Percentage of Subjects With Dengue Virus Antibody IgG Positive Result (ELISA) at First Visit (Indicative of Past DENV Infection), by Study Site and Age Category.
Description: The percentage of subjects with Dengue Virus antibody IgG positive result (ELISA) was expressed as percentage of subjects = (n [number of subjects with at least one event reported during the study period]/N [number of subjects in the population]) X 100. The 95% Wald CI was calculated. Clustering effect was not retained because equal or less than 1. Ages categories were defined as follows: "6 months -<12 Months" = from the 6 Months birthday up to and including the day before the 1st year birthday, and the next "n-p Years" categories = from the nth Year birthday up to and including the day before the (p+1)th Year birthday. Analysis was not summarized for confirmed and probable dengue cases, separately as there were no probable cases reported in the study.
Time Frame: At Day 0
Population: Analysis was performed on the According-to-Protocol cohort that included all evaluable subjects from Mexico (1-4 years age) and the Philippines (6-12 months), i.e. subjects who met all eligibility criteria, complying with the procedures defined in the protocol and for whom data of at least one follow-up contact were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Total Group
Number analyzed (Participants) | 59
Percentage of subjects
  Mexico- 1-4 years: number analyzed (Participants) | 47
  Mexico- 1-4 years | 6.4 [2.1 to 18.0]
  Philippines- 6 months -12 months: number analyzed (Participants) | 12
  Philippines- 6 months -12 months | 8.3 [1.2 to 41.3]

8. Secondary Outcome: Number of Suspected Dengue Cases With Temperature and Any Symptom From First and Returned Visits
Description: The following characteristics were summarized for each category of dengue cases (Virologically confirmed, probable, other SDC): Temperature at first visit: <37.5, ≥37.5, >38, >38.5, >39 °C and Clinical symptoms at onset, from first and returned visits. The results are presented for the virologically confirmed cases (VDC) and the other SDC (oSDC), no probable cases being reported in the study.
Time Frame: From Day 0 to Month 24 (study end)
Population: Analysis was performed on the According-to-Protocol cohort that included all evaluable subjects, i.e. subjects who met all eligibility criteria, complying with the procedures defined in the protocol, for whom data of at least one follow-up contact were available and who were defined as suspected dengue cases.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 27
Participants
  Temperature <37.5 °C VDC: number analyzed (Participants) | 9
  Temperature <37.5 °C VDC | 5
  Temperature ≥37.5 °C VDC: number analyzed (Participants) | 9
  Temperature ≥37.5 °C VDC | 4
  Temperature >38.0 °C VDC: number analyzed (Participants) | 9
  Temperature >38.0 °C VDC | 4
  Temperature >38.5 °C VDC: number analyzed (Participants) | 9
  Temperature >38.5 °C VDC | 1
  Temperature >39.0 °C VDC: number analyzed (Participants) | 9
  Temperature >39.0 °C VDC | 0
  At least one main sign VDC: number analyzed (Participants) | 9
  At least one main sign VDC | 9
  Fever VDC: number analyzed (Participants) | 9
  Fever VDC | 9
  Headache VDC: number analyzed (Participants) | 9
  Headache VDC | 7
  Retroorbital pain [eye pain] VDC: number analyzed (Participants) | 9
  Retroorbital pain [eye pain] VDC | 6
  Myalgia VDC: number analyzed (Participants) | 9
  Myalgia VDC | 5
  Join pain VDC: number analyzed (Participants) | 9
  Join pain VDC | 3
  Chills VDC: number analyzed (Participants) | 9
  Chills VDC | 2
  Rash VDC: number analyzed (Participants) | 9
  Rash VDC | 1
  Itching VDC: number analyzed (Participants) | 9
  Itching VDC | 1
  At least one digestive symptom VDC: number analyzed (Participants) | 9
  At least one digestive symptom VDC | 5
  Abdominal pain VDC: number analyzed (Participants) | 9
  Abdominal pain VDC | 5
  Nausea or vomiting VDC: number analyzed (Participants) | 9
  Nausea or vomiting VDC | 4
  Diarrhea VDC: number analyzed (Participants) | 9
  Diarrhea VDC | 2
  At least one respiratory symptom VDC: number analyzed (Participants) | 9
  At least one respiratory symptom VDC | 5
  Cough VDC: number analyzed (Participants) | 9
  Cough VDC | 4
  Nasal Congestion VDC: number analyzed (Participants) | 9
  Nasal Congestion VDC | 2
  Sore throat VDC: number analyzed (Participants) | 9
  Sore throat VDC | 1
  Dyspnea VDC: number analyzed (Participants) | 9
  Dyspnea VDC | 0
  At least one hemorrhagic manifestation VDC: number analyzed (Participants) | 9
  At least one hemorrhagic manifestation VDC | 1
  Petechia VDC: number analyzed (Participants) | 9
  Petechia VDC | 1
  Purpura/ecchymosis VDC: number analyzed (Participants) | 9
  Purpura/ecchymosis VDC | 0
  Hematemesis [vomiting of blood] VDC: number analyzed (Participants) | 9
  Hematemesis [vomiting of blood] VDC | 0
  Melena/hematochezia [blood in stool] VDC: number analyzed (Participants) | 9
  Melena/hematochezia [blood in stool] VDC | 0
  Gingival bleeding VDC: number analyzed (Participants) | 9
  Gingival bleeding VDC | 0
  Epistaxis VDC: number analyzed (Participants) | 9
  Epistaxis VDC | 0
  Urinary tract bleeding VDC: number analyzed (Participants) | 9
  Urinary tract bleeding VDC | 0
  Unusual vaginal bleeding VDC: number analyzed (Participants) | 9
  Unusual vaginal bleeding VDC | 0
  At least one other signs VDC: number analyzed (Participants) | 9
  At least one other signs VDC | 6
  Pallor or cool skin VDC: number analyzed (Participants) | 9
  Pallor or cool skin VDC | 0
  Conjunctivis VDC: number analyzed (Participants) | 9
  Conjunctivis VDC | 1
  Jaundice VDC: number analyzed (Participants) | 9
  Jaundice VDC | 0
  Convulsion or coma VDC: number analyzed (Participants) | 9
  Convulsion or coma VDC | 0
  Lethargy or restlessness VDC: number analyzed (Participants) | 9
  Lethargy or restlessness VDC | 0
  Clinical fluid accumulation VDC: number analyzed (Participants) | 9
  Clinical fluid accumulation VDC | 1
  Dizziness VDC: number analyzed (Participants) | 9
  Dizziness VDC | 1
  Thoracic pain VDC: number analyzed (Participants) | 9
  Thoracic pain VDC | 0
  Other VDC: number analyzed (Participants) | 9
  Other VDC | 6
  Temperature <37.5 °C oSDC: number analyzed (Participants) | 18
  Temperature <37.5 °C oSDC | 15
  Temperature ≥37.5 °C oSDC: number analyzed (Participants) | 18
  Temperature ≥37.5 °C oSDC | 3
  Temperature >38.0 °C oSDC: number analyzed (Participants) | 18
  Temperature >38.0 °C oSDC | 2
  Temperature >38.5 °C oSDC: number analyzed (Participants) | 18
  Temperature >38.5 °C oSDC | 0
  Temperature >39.0 °C oSDC: number analyzed (Participants) | 18
  Temperature >39.0 °C oSDC | 0
  At least one main sign oSDC: number analyzed (Participants) | 18
  At least one main sign oSDC | 18
  Fever oSDC: number analyzed (Participants) | 18
  Fever oSDC | 18
  Headache oSDC: number analyzed (Participants) | 18
  Headache oSDC | 15
  Retroorbital pain [eye pain] oSDC: number analyzed (Participants) | 18
  Retroorbital pain [eye pain] oSDC | 9
  Myalgia oSDC: number analyzed (Participants) | 18
  Myalgia oSDC | 11
  Join pain oSDC: number analyzed (Participants) | 18
  Join pain oSDC | 8
  Chills oSDC: number analyzed (Participants) | 18
  Chills oSDC | 2
  Rash oSDC: number analyzed (Participants) | 18
  Rash oSDC | 4
  Itching oSDC: number analyzed (Participants) | 18
  Itching oSDC | 1
  At least one digestive symptom oSDC: number analyzed (Participants) | 18
  At least one digestive symptom oSDC | 12
  Abdominal pain oSDC: number analyzed (Participants) | 18
  Abdominal pain oSDC | 8
  Nausea or vomiting oSDC: number analyzed (Participants) | 18
  Nausea or vomiting oSDC | 11
  Diarrhea oSDC: number analyzed (Participants) | 18
  Diarrhea oSDC | 2
  At least one respiratory symptom oSDC: number analyzed (Participants) | 18
  At least one respiratory symptom oSDC | 11
  Cough oSDC: number analyzed (Participants) | 18
  Cough oSDC | 8
  Nasal Congestion oSDC: number analyzed (Participants) | 18
  Nasal Congestion oSDC | 6
  Sore throat oSDC: number analyzed (Participants) | 18
  Sore throat oSDC | 2
  Dyspnea oSDC: number analyzed (Participants) | 18
  Dyspnea oSDC | 1
  At least one hemorrhagic manifestation oSDC: number analyzed (Participants) | 18
  At least one hemorrhagic manifestation oSDC | 1
  Petechia oSDC: number analyzed (Participants) | 18
  Petechia oSDC | 0
  Purpura/ecchymosis oSDC: number analyzed (Participants) | 18
  Purpura/ecchymosis oSDC | 0
  Hematemesis [vomiting of blood] oSDC: number analyzed (Participants) | 18
  Hematemesis [vomiting of blood] oSDC | 0
  Melena/hematochezia [blood in stool] oSDC: number analyzed (Participants) | 18
  Melena/hematochezia [blood in stool] oSDC | 0
  Gingival bleeding oSDC: number analyzed (Participants) | 18
  Gingival bleeding oSDC | 1
  Epistaxis oSDC: number analyzed (Participants) | 18
  Epistaxis oSDC | 1
  Urinary tract bleeding oSDC: number analyzed (Participants) | 18
  Urinary tract bleeding oSDC | 0
  Unusual vaginal bleeding oSDC: number analyzed (Participants) | 18
  Unusual vaginal bleeding oSDC | 0
  At least one other signs oSDC: number analyzed (Participants) | 18
  At least one other signs oSDC | 10
  Pallor or cool skin oSDC: number analyzed (Participants) | 18
  Pallor or cool skin oSDC | 0
  Conjunctivis oSDC: number analyzed (Participants) | 18
  Conjunctivis oSDC | 1
  Jaundice oSDC: number analyzed (Participants) | 18
  Jaundice oSDC | 0
  Convulsion or coma oSDC: number analyzed (Participants) | 18
  Convulsion or coma oSDC | 0
  Lethargy or restlessness oSDC: number analyzed (Participants) | 18
  Lethargy or restlessness oSDC | 2
  Clinical fluid accumulation oSDC: number analyzed (Participants) | 18
  Clinical fluid accumulation oSDC | 0
  Dizziness oSDC: number analyzed (Participants) | 18
  Dizziness oSDC | 2
  Thoracic pain oSDC: number analyzed (Participants) | 18
  Thoracic pain oSDC | 0
  Other oSDC: number analyzed (Participants) | 18
  Other oSDC | 7

9. Secondary Outcome: Number of Suspected Dengue Cases With Severity Criteria Characteristics
Description: The clinical classification of the suspected dengue cases were distributed among following categories: Subject hospitalized during suspected dengue episode; OR At least 1 WHO 2009 warning signs: i.e. Abdominal pain or tenderness, Persistent vomiting, Clinical fluid accumulation, Mucosal bleed, Liver enlargement, Increase in HCT concurrent with rapid decrease in platelet count, Lethargy and restlessness; OR At least 1 WHO 2009 criteria for severe dengue: i.e. Severe Plasma Leakage leading to Shock, Fluid accumulation with respiratory distress, Severe Bleeding, Severe organ involvement; Liver: Aspartate transaminase or Alanine transferase ≥ 1000 International Unit/Liter, Central nervous system: impaired consciousness, Failure of heart and other organs; OR Most likely diagnosis for an episode of defined illnesses [investigator opinion]. The following characteristics were summarized for Virologically confirmed cases (VDC) and other SDC (oSDC), no probable cases being reported.
Time Frame: From Day 0 to Month 24 (study end)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 27
Participants
  Subject hospitalized VDC: number analyzed (Participants) | 9
  Subject hospitalized VDC | 0
  At least 1 WHO 2009 warning signs VDC: number analyzed (Participants) | 9
  At least 1 WHO 2009 warning signs VDC | 5
  At least 1 WHO 2009 severe dengue criteria VDC: number analyzed (Participants) | 9
  At least 1 WHO 2009 severe dengue criteria VDC | 0
  Most likely diagnosis: Dengue VDC: number analyzed (Participants) | 9
  Most likely diagnosis: Dengue VDC | 7
  Most likely diagnosis: Chikungunya VDC: number analyzed (Participants) | 9
  Most likely diagnosis: Chikungunya VDC | 0
  Most likely diagnosis: Influenza VDC: number analyzed (Participants) | 9
  Most likely diagnosis: Influenza VDC | 0
  Most likely diagnosis: Malaria VDC: number analyzed (Participants) | 9
  Most likely diagnosis: Malaria VDC | 0
  Most likely diagnosis: Leptospirosis VDC: number analyzed (Participants) | 9
  Most likely diagnosis: Leptospirosis VDC | 0
  Most likely diagnosis: Rota/enteric infection VDC: number analyzed (Participants) | 9
  Most likely diagnosis: Rota/enteric infection VDC | 0
  Most likely diagnosis: other infection disease VDC: number analyzed (Participants) | 9
  Most likely diagnosis: other infection disease VDC | 2
  Most likely diagnosis: non-infectious disease VDC: number analyzed (Participants) | 9
  Most likely diagnosis: non-infectious disease VDC | 0
  Subject hospitalized oSDC: number analyzed (Participants) | 18
  Subject hospitalized oSDC | 0
  At least 1 WHO 2009 warning signs oSDC: number analyzed (Participants) | 18
  At least 1 WHO 2009 warning signs oSDC | 1
  At least 1 WHO 2009 severe dengue criteria oSDC: number analyzed (Participants) | 18
  At least 1 WHO 2009 severe dengue criteria oSDC | 0
  Most likely diagnosis: Dengue oSDC: number analyzed (Participants) | 18
  Most likely diagnosis: Dengue oSDC | 2
  Most likely diagnosis: Chikungunya oSDC: number analyzed (Participants) | 18
  Most likely diagnosis: Chikungunya oSDC | 0
  Most likely diagnosis: Influenza oSDC: number analyzed (Participants) | 18
  Most likely diagnosis: Influenza oSDC | 2
  Most likely diagnosis: Malaria oSDC: number analyzed (Participants) | 18
  Most likely diagnosis: Malaria oSDC | 0
  Most likely diagnosis: Leptospirosis oSDC: number analyzed (Participants) | 18
  Most likely diagnosis: Leptospirosis oSDC | 0
  Most likely diagnosis: Rota/enteric infection oSDC: number analyzed (Participants) | 18
  Most likely diagnosis: Rota/enteric infection oSDC | 0
  Most likely diagnosis: other infection oSDC: number analyzed (Participants) | 18
  Most likely diagnosis: other infection oSDC | 18
  Most likely diagnosis: non-infectious disease oSDC: number analyzed (Participants) | 18
  Most likely diagnosis: non-infectious disease oSDC | 0

10. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Related to a Study Procedure
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject..
Time Frame: From Day 0 to Month 24 (study end)
Population: Analysis was performed on the Total cohort that included all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Group
Number analyzed (Participants) | 850
Participants | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from Day 0 to Month 24 (study end).
Description: Other Adverse Events were not collected in this study.
Arm/Group | Total Group
All-Cause Mortality (participants affected / at risk) | 1/850
Serious Adverse Events (participants affected / at risk) | 0/850
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Analyses by season/year, age, gender, serotype and dengue serological status at beginning of analysis period were not performed due to low number of virologically confirmed or probable symptomatic dengue infection reported during the study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT02766088/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT02766088/SAP_001.pdf